CLINICAL TRIAL: NCT05508672
Title: Community-Centered eHealth Smoking Cessation Intervention Based on the "Smoking Rationalization Beliefs" Framework for Chinese Male Smokers
Brief Title: Community-Centered eHealth Smoking Cessation Intervention(CCeSCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke Kunshan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22KDKUF016
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Smoking Cessation; Lifestyle, Healthy
Keywords: Smoking Cessation; Disease control and prevention; Health management; Effectiveness evaluation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-Centered eHealth Smoking Cessation Intervention (CCeSCI) group (Experimental): The intervention group will receive Community-Centered eHealth Smoking Cessation Intervention(CCeSCI).
  Interventions: Other: Community-Centered eHealth Smoking Cessation Intervention (CCeSCI)
- Traditional "smoking is harmful" education group (Active Comparator): The control group to receive the traditional "smoking is harmful" education.
  Interventions: Other: Traditional "smoking is harmful" education

INTERVENTIONS:
Other: Community-Centered eHealth Smoking Cessation Intervention (CCeSCI) — We will equip CCeSCI with both core eHealth features and provider-side intervention. Patients assigned to the intervention group will receive a series of online interactive and personalization technologies, including an algorithm-based video curriculum with auto-texting, backstage monitoring system etc. Besides, the patients will also have the face-to-face meetings with community health workers. Provider-side intervention includes training for community workers, WeChat group discussion, and performance-based incentives. The training aims to provide essential skills for community workers so that they can provide face-to-face meetings with smokers during the first 3 months of quitting to prevent or revert relapse in a timely and proactive manner.
  Arms: Community-Centered eHealth Smoking Cessation Intervention (CCeSCI) group
Other: Traditional "smoking is harmful" education — In the control group, the participants will receive traditional "smoking is harmful" education video, which is recorded by the clinical physicians.
  Arms: Traditional "smoking is harmful" education group

SUMMARY:
Recent findings regarding why Chinese male smokers are reluctant to quit have offered insight for a possible new solution. Consistent with the Cognitive Dissonance Theory, "smoking rationalization beliefs" are a set of beliefs by smokers to rationalize their smoking behavior and avoid quitting. These beliefs have been well studied by global researchers, and a "smoking rationalization beliefs" scale was recently developed and validated for Chinese male smokers. The six dimensions of these beliefs are: smoking functional beliefs, risk generalization beliefs, social acceptability beliefs, safe smoking beliefs, self-exempting beliefs, and quitting is harmful beliefs. Studies on smoking rationalization in China have primarily been observational. Investigators propose to develop a Community-Centered eHealth Smoking Cessation Intervention (CCeSCI). The trinity of CCeSCI are the triangular unity of "smoking rationalization beliefs" framework, the non-physician community workers, and the eHealth technologies. The latter two were previously proven effective in interventional studies (including three conducted by the PI) but not yet widely used in smoking cessation. With the adoption of smoking rationalization beliefs framework aiming to address the cognitive causes of phycological addition to smoking and supported by the community-based behavioral interventions and the use of eHealth, CCeSCI is designed to overcome previous challenges with the principles of people-centeredness, convenience, and personalization.

DETAILED DESCRIPTION:
Investigators will firstly evaluate the feasibility of CCeSCI. Once CCeSCI is ready to deploy, investigators will recruit 60 smokers (male, 25-64 years old) in two communities in Qingpu to conduct a pilot non-blinded randomized controlled trial. They will be randomized in a 1:1 ratio into either the intervention group to receive CCeSCI or the control group to receive the traditional "smoking is harmful" education video. Investigators will also use qualitative research methods (one on one interviews) to conduct process evaluations at 4th, 8th, and 12th weeks according to the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework. At the end of the 12th week after the participants joined the RCT, saliva samples will be collected by community workers and quitting outcomes will be biochemically verified by a third party lab.

ELIGIBILITY:
Inclusion Criteria:

1. Male, current cigarette smokers who are willing to quit
2. Citizens who currently reside in Qingpu District, Shanghai, China
3. Age 25-64
4. Smoking index greater than or equal to 100 (smoking index = average number of cigarettes smoked per day × years of smoking)
5. Able to understand mandarin Chinese
6. Willing to provide informed consent to participate in the study

Exclusion Criteria:

1. Ever or currently on pharmacologic treatments, including various forms of NRT formulations such as gum, transdermal patch, nasal spray, oral inhaler, lozenge, Bupropion, Varenicline and newly emerged precision medicine
2. Currently participating in other individual-based cessation program(s), such as psychological counseling, behavioral therapy etc.
3. Currently under treatment of life-threatening medical conditions or critically ill
4. Unable to make commitment of a consecutive 4-hour video viewing
5. Plan to move out of the community in the next 3 month

Ages: 25 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The eligible participants are male smokers.
Enrollment: 60 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Biochemically verified continuous smoking abstinence at 3 month | 3 month
  Investigators will use cotinine to measure the smoking abstinence. Cotinine is a good biomarker for nicotine with a longer half-life (16-18h), and lab test for saliva is highly sensitive, convenient, and cost-effective. measured by cotinine saliva tests (<10ng•mL-1)

SECONDARY OUTCOMES:
Fagerstrom Test For Nicotine Dependence (FTND) Score | Change from baseline to 3-month follow up
  Investigators will use the Fagerström Test for Nicotine Dependence as a standard instrument for assessing the intensity of physical addiction to nicotine. In scoring the Fagerstrom Test for Nicotine Dependence, the three yes/no items are scored 0 (no) and 1 (yes). The three multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. A higher score means more dependence on nicotine.
Patient Health Questionnaire-9 | Change from baseline to 3-month follow up
  Investigators will use PHQ-9 as a 9-question instrument to screen for depression. The scale ranges from 0 to 27. Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe, and severe depression, respectively. Higher score indicates severe depression
Self-reported 7-day point smoking status | 3-month follow up
  self-reported 7-day point prevalence of abstinence (not even a puff of smoke, for the last 7 days) at 3 months
Self-reported continuous abstinence at 3 month | 3-month follow up
  not even a puff of smoke, for the last 3 months
Self-reported average number of cigarettes | Change from baseline to 3-month follow up
  Investigators will count the number of cigarettes at 3 month
Smoking Rationalization Scale | Change from baseline to 3-month follow up
  Investigators will use Smoking Rationalization Scale to measure smokers' thoughts about smoking. The scale comprised 26 items (e.g., "Smoking is good for inspiration and active thinking.") and was divided into 6 dimensions including smoking functional beliefs, risk generalization beliefs, social acceptability beliefs, safe smoking beliefs, self-exempting beliefs and quitting is harmful beliefs. Participants responded on a 5-point Likert scale (1 = completely disagree, 5 = completely agree). Higher scores indicated a higher level of smoking rationalization beliefs.
Questionnaire about community health workers' Knowledge, Attitude and Practices (KAP) | 3-month follow up
  The knowledge, attitude, and practices (KAPs) survey provides a design to evaluate existing programs and to identify effective strategies for behavior change in society. The first section was related to knowledge, and this section had some questions where 1 point was assigned to the correct answer and 0 points were assigned to the wrong answer. A higher score demonstrated good knowledge. The second section was on attitude and had some questions on a 5-point Likert scale as strongly disagree = 1, disagree = 2, uncertain = 3, agree = 4, and strongly agree = 5. A higher score demonstrated a good attitude. The last part of the questionnaire was composed of questions related to the practice, and each question was scored as "yes" (1-point), "no" (0-point), and "sometimes" (0-point). A higher score indicated good practice.
Weight in kilograms | Change from baseline to 3-month follow up
  Investigators will measure the participants' heights
Blood Pressure | Change from baseline to 3-month follow up
  Investigators will measure the participants' both systolic and diastolic blood pressure
Waist Circumference | Change from baseline to 3-month follow up
  Investigators will measure the waist circumference of the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Qingpu Patriotic Hygiene and Health Promotion Guidance Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The investigators will not share the individual participant data. But de-identified data is available upon request.

REFERENCES:
- [Background] GBD 2015 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 79 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1659-1724. doi: 10.1016/S0140-6736(16)31679-8. PMID 27733284
- [Background] Wang L, Shen Y, Jiang Y, Yang Y. [Investigation and analysis on current status of smoking cessation clinics in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2015 Sep;36(9):917-20. Chinese. PMID 26814853
- [Background] Wang J, Xie L, Jiang Y, Li Q. Conclusions and impacts of U.S. Surgeon General' s Reports on smoking and tobacco use. Chinese Journal of Health Education 2012;28(7):591-593+601. DOI: 10.16168/j.cnki.issn.1002-9982.2012.07.019.
- [Background] Huang X, Fu W, Zhang H, Li H, Li X, Yang Y, Wang F, Gao J, Zheng P, Fu H, Chapman S, Ding D. Why are male Chinese smokers unwilling to quit? A multicentre cross-sectional study on smoking rationalisation and intention to quit. BMJ Open. 2019 Feb 19;9(2):e025285. doi: 10.1136/bmjopen-2018-025285. PMID 30782929
- [Background] Fotuhi O, Fong GT, Zanna MP, Borland R, Yong HH, Cummings KM. Patterns of cognitive dissonance-reducing beliefs among smokers: a longitudinal analysis from the International Tobacco Control (ITC) Four Country Survey. Tob Control. 2013 Jan;22(1):52-8. doi: 10.1136/tobaccocontrol-2011-050139. Epub 2012 Jan 3. PMID 22218426
- [Background] Huang X, Fu W, Zhang H, Li H, Li X, Yang Y, Wang F, Gao J, Zheng P, Fu H, Ding D, Chapman S. Development and validation of a smoking rationalization scale for male smokers in China. J Health Psychol. 2020 Mar;25(4):472-489. doi: 10.1177/1359105317720276. Epub 2017 Jul 20. PMID 28810494
- [Background] Chen S, Gong E, Kazi DS, Gates AB, Bai R, Fu H, Peng W, De La Cruz G, Chen L, Liu X, Su Q, Girerd N, Karaye KM, Alhabib KF, Yan LL, Schwalm JD. Using Mobile Health Intervention to Improve Secondary Prevention of Coronary Heart Diseases in China: Mixed-Methods Feasibility Study. JMIR Mhealth Uhealth. 2018 Jan 25;6(1):e9. doi: 10.2196/mhealth.7849. PMID 29371178
- [Background] Gong E, Gu W, Luo E, Tan L, Donovan J, Sun C, Yang Y, Zang L, Bao P, Yan LL. Development and Local Contextualization of Mobile Health Messages for Enhancing Disease Management Among Community-Dwelling Stroke Patients in Rural China: Multimethod Study. JMIR Mhealth Uhealth. 2019 Dec 17;7(12):e15758. doi: 10.2196/15758. PMID 31845901
- [Background] Gong E, Sun L, Long Q, Xu H, Gu W, Bettger JP, Tan J, Ma J, Jafar TH, Oldenburg B, Yan LL. The Implementation of a Primary Care-Based Integrated Mobile Health Intervention for Stroke Management in Rural China: Mixed-Methods Process Evaluation. Front Public Health. 2021 Nov 17;9:774907. doi: 10.3389/fpubh.2021.774907. eCollection 2021. PMID 34869187
- [Background] Ni Z, Liu C, Wu B, Yang Q, Douglas C, Shaw RJ. An mHealth intervention to improve medication adherence among patients with coronary heart disease in China: Development of an intervention. Int J Nurs Sci. 2018 Sep 8;5(4):322-330. doi: 10.1016/j.ijnss.2018.09.003. eCollection 2018 Oct 10. PMID 31406843
- [Background] Yan LL, Gong E, Gu W, Turner EL, Gallis JA, Zhou Y, Li Z, McCormack KE, Xu LQ, Bettger JP, Tang S, Wang Y, Oldenburg B. Effectiveness of a primary care-based integrated mobile health intervention for stroke management in rural China (SINEMA): A cluster-randomized controlled trial. PLoS Med. 2021 Apr 28;18(4):e1003582. doi: 10.1371/journal.pmed.1003582. eCollection 2021 Apr. PMID 33909607
- [Background] Tian M, Ajay VS, Dunzhu D, Hameed SS, Li X, Liu Z, Li C, Chen H, Cho K, Li R, Zhao X, Jindal D, Rawal I, Ali MK, Peterson ED, Ji J, Amarchand R, Krishnan A, Tandon N, Xu LQ, Wu Y, Prabhakaran D, Yan LL. A Cluster-Randomized, Controlled Trial of a Simplified Multifaceted Management Program for Individuals at High Cardiovascular Risk (SimCard Trial) in Rural Tibet, China, and Haryana, India. Circulation. 2015 Sep 1;132(9):815-24. doi: 10.1161/CIRCULATIONAHA.115.015373. Epub 2015 Jul 17. PMID 26187183